CLINICAL TRIAL: NCT06719401
Title: Comparing Foot and Hand Cardiopulmonary Resuscitation: a Non- Inferiority, Crossover, Randomised Controlled Simulation Study
Brief Title: Comparing Foot and Hand CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Keon Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B-2205-758-302
Record Dates: First submitted 2024-11-24; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Arrest (CA); Simulation Training
Keywords: foot CPR; simulation study
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- F-H Group (Other): Participants in this group perform training and testing using the foot chest compression (FCC) method first, followed by training and testing using the hand chest compression (HCC) method.
  Interventions: Other: Foot Chest Compression; Other: Hand Chest Compression
- H-F Group (Other): Participants in this group perform training and testing using the hand chest compression (HCC) method first, followed by training and testing using the foot chest compression (FCC) method.
  Interventions: Other: Foot Chest Compression; Other: Hand Chest Compression

INTERVENTIONS:
Other: Foot Chest Compression — Foot chest compression is an alternative cardiopulmonary resuscitation (CPR) technique where the rescuer uses one foot to perform compressions on the chest instead of their hands. The heel of the foot is placed on the lower half of the sternum, with the foot parallel to the sternum to ensure effective pressure. The opposite foot provides stability by being positioned beside the patient.
Other: Hand Chest Compression — Hand chest compression is the conventional method of performing chest compressions during CPR. It involves the use of both hands, with one hand placed over the other on the lower half of the sternum. The rescuer positions their body directly over the patient, using the weight of their upper body to deliver compressions of 50-60 mm depth at a rate of 100-120 compressions per minute. Proper technique includes full chest recoil between compressions, maintaining a straight arm posture, and avoiding pressure on the xiphoid process to minimize injury risks. This method adheres to the 2020 AHA guidelines for high-quality CPR.

SUMMARY:
The goal of this simulation study is to evaluate whether chest compression using the foot is comparable to chest compression using the hand during cardiopulmonary resuscitation in trained participants. This study aims to compare the effectiveness of hand chest compression (HCC) with foot chest compression (FCC) and investigate differences in their efficacy based on rescuer characteristics through subgroup analysis. It is designed as a simulation study to assess the efficacy of the FCC method as an alternative to HCC without exposing patients to risk.

DETAILED DESCRIPTION:
Study Design and Setting This is a prospective, crossover, non-inferiority, randomised controlled trial. We hypothesise that the FCC method is not inferior to the existing HCC method regarding depth, rate, and chest compression position. The study is approved by the Institutional Review Board (IRB) of Seoul National University Bundang Hospital (B-2205-758-302).

The primary outcomes of this study are the mean chest compression depth (mm) and mean chest compression rate (n/min) for 2 minutes. The secondary outcomes are the proportions of adequate compression depth (%), adequate compression rate (%), adequate compression depth and rate (%), correct chest compression position (%), and compression with full release (%). According to the 2020 AHA Cardiopulmonary Resuscitation and Emergency Cardiovascular Care guidelines, adequate compression depth is defined as a compression of 50-60 mm, and adequate compression rate is defined as a rate of 100-120 compressions per minute. The correct chest compression position is measured using a manikin simulator to ensure that the lower half of the sternum is compressed accurately. If the location of chest compression is incorrect, the chest movement tilts instead of moving horizontally, and this is deemed as an incorrect compression.

Participant Enrollment Participants are recruited through a poster on the information board of a university, following IRB approval. The inclusion criteria for participants are adults aged over 18 years who are certified as AHA Basic Life Support (BLS) providers or have undergone equivalent BLS training. Applicants who meet the following criteria are excluded because they are judged unable to perform adequate chest compressions: (1) physical or cognitive disabilities and (2) musculoskeletal injuries, such as limb injuries. Additionally, as the study is conducted during the COVID-19 pandemic, individuals diagnosed with COVID-19, under quarantine, or experiencing fever or respiratory symptoms suspected to be COVID-19 are excluded.

The purpose of the study is explained to participants who meet the inclusion criteria, including their right to withdraw consent at any time. Participants then complete a written informed consent form to participate in the study.

Simulation Design Participants attend a brief educational session covering the theoretical content of chest compressions, including the importance of compression position, depth, rate, and full release. Education is provided following the 2020 AHA Cardiopulmonary Resuscitation and Emergency Cardiovascular Care guidelines. Additionally, the session includes an explanation of chest compression methods using both hands and feet.

After the educational session, participants are divided into a foot-hand group (F-H group) and a hand-foot group (H-F group) according to whether FCC or HCC is performed first, through random allocation. Participants are then moved to independent rooms (Room A for the F-H group and Room B for the H-F group).

This study uses a crossover design. Participants in the F-H group first perform training and testing using the FCC method and then perform training and testing using the HCC method, while participants in the H-F group follow the opposite order.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Certified AHA basic life support provider or undergone equivalent BLS training

Exclusion Criteria:

* Unable to perform adequate chest compressions due to:

  1. physical or cognitive disabilities
  2. musculoskeletal injuries, such as limb injuries.
* Diagnosed with COVID-19 and quarantined
* Complained of fever or respiratory symptoms suspected to be COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
mean chest compression depth | 1 week after completion of simulation.
  The mean chest compression depth refers to the average depth (mm) achieved during chest compressions for 2 minutes.

SECONDARY OUTCOMES:
adequate compression depth | 1 week after completion of simulation.
  Adequate compression depth is defined as a compression of 50-60 mm, and in this study the percentage of adequate compression depth achieved during a 2 minute period will be calculated.
adequate compression rate | 1 week after completion of simulation.
  Adequate compression rate is defined as a compression rate of 100-120/min, and in this study the percentage of adequate compression rate achieved during a 2 minute period will be calculated.
adequate compression depth and rate | 1 week after completion of simulation.
  The percentage of compressions achieving both adequate compression depth and rate will be obtained.
correct chest compression position | 1 week after completion of simulation.
  The correct chest compression position will be measured using a manikin simulator to ensure that the lower half of the sternum was compressed accurately. The percentage of correct chest compression position will be obtained.
compression with full release | 1 week after completion of simulation.
  The percentage of compression with full release will be obtained using the manikin simulator.
mean chest compression rate | 1 week after completion of simulation.
  The mean chest compression rate represents the average number of compressions delivered per minute (n/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univeristy Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trenkamp RH, Perez FJ. Heel compressions quadruple the number of bystanders who can perform chest compressions for 10 minutes. Am J Emerg Med. 2015 Oct;33(10):1449-53. doi: 10.1016/j.ajem.2015.06.070. Epub 2015 Jul 6. PMID 26298049
- [Background] Hung TY, Wen CS, Yu SH, Chen YC, Chen HL, Chen WL, Wu CC, Su YC, Lin CL, Hu SC, Lin T. A comparative analysis of aerosol exposure and prevention strategies in bystander, pre-hospital, and inpatient cardiopulmonary resuscitation using simulation manikins. Sci Rep. 2023 Aug 2;13(1):12552. doi: 10.1038/s41598-023-39726-x. PMID 37532861
- [Background] Bylow H, Karlsson T, Claesson A, Lepp M, Lindqvist J, Herlitz J. Self-learning training versus instructor-led training for basic life support: A cluster randomised trial. Resuscitation. 2019 Jun;139:122-132. doi: 10.1016/j.resuscitation.2019.03.026. Epub 2019 Mar 26. PMID 30926451
- [Background] Wong MF, Ho MP. Leg-heel chest compression as an alternative for medical professionals in times of COVID-19. Am J Emerg Med. 2022 Jul;57:222. doi: 10.1016/j.ajem.2022.02.026. Epub 2022 Feb 19. No abstract available. PMID 35219559
- [Background] Peberdy MA, Silver A, Ornato JP. Effect of caregiver gender, age, and feedback prompts on chest compression rate and depth. Resuscitation. 2009 Oct;80(10):1169-74. doi: 10.1016/j.resuscitation.2009.07.003. Epub 2009 Aug 11. PMID 19674826
- [Background] Kherbeche H, Exer N, Schuhwerk W, Ummenhofer W, Osterwalder J. Chest compression using the foot or hand method: a prospective, randomized, controlled manikin study with school children. Eur J Emerg Med. 2017 Aug;24(4):262-267. doi: 10.1097/MEJ.0000000000000335. PMID 26485692
- [Background] Bae GE, Choi A, Beom JH, Kim MJ, Chung HS, Min IK, Chung SP, Kim JH. Correlation between real-time heart rate and fatigue in chest compression providers during cardiopulmonary resuscitation: A simulation-based interventional study. Medicine (Baltimore). 2021 Apr 23;100(16):e25425. doi: 10.1097/MD.0000000000025425. PMID 33879672